CLINICAL TRIAL: NCT05784155
Title: A Randomized, Open-label, Multiple-dose, Crossover Phase I Clinical Trial to Compare the Safety, Pharmacokinetics and Pharmacodynamics After Oral Administration of JW0302 to C2206 in Healthy Adult Subjects
Brief Title: To Evaluate the PK, PD, Safety and Drug Tolerance of JW0302 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: JW22106
Record Dates: First submitted 2023-03-01; First posted 2023-03-24 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: A randomized, open, single-dose, 2x2 crossover-design clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): Test Drug for Period I Reference Drug for Period II
  Interventions: Drug: Test Drug(JW0302) or Reference Drug(C2206)
- Group 2 (Other): Reference Drug for Period I Test Drug for Period II
  Interventions: Drug: Test Drug(JW0302) or Reference Drug(C2206)

INTERVENTIONS:
Drug: Test Drug(JW0302) or Reference Drug(C2206) — Test Drug: single administration of JW0302 Reference Drug: single administration of C2206
  Tablet, Oral, QD for 1 Days, Washout period is more than 14 days after administration

SUMMARY:
1. To evaluate the pharmacokinetic and pharmacodynamics characteristics after administration of Reference Drug or Test Drug in healthy volunteers under fasting conditions
2. To evaluate the safety and drug tolerance after administration of Reference Drug or Test Drug in healthy volunteers under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Subjects does not meet the Inclusion Criteria

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
AUCτ, SS(Area under the plasma drug concentration-time curve within a dosing interval at steady state) | up to 24 hours
  Evaluation PK for JW0302 and C2206 after multiple dose
Percent decrease from baseline in integrated gastric acidity for 24-hour interval after 7th dose | Baseline versus Multiple dose during 7 days
  Evaluation PD for ambulatory 24hr pH monitor

CONTACTS AND LOCATIONS:
Overall Officials: SeungHwan Lee, PI, Principal Investigator — Clinical Trial Center, Seoul National University Hospital
Locations (1):
- Clinical Trial Center, Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No